CLINICAL TRIAL: NCT03846141
Title: Hydrogen Inhalation for Health and Exercise Performance
Acronym: HIHEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UniversityNSFSandPE
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Exercise Performance
MeSH Terms: interventions — Hydrogen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Room air for inhalation
  Interventions: Other: Placebo
- Hydrogen (Experimental): Hydrogen (4%) for inhalation
  Interventions: Other: Hydrogen

INTERVENTIONS:
Other: Placebo — Inhalation of room air for 20 min per day during 7 days
  Arms: Placebo
Other: Hydrogen — Inhalation of 4% hydrogen for 20 min per day during 7 days
  Arms: Hydrogen

SUMMARY:
In this randomized double-blind, placebo-controlled, crossover pilot trial, we evaluated the effects of 7-day H2 inhalation on exercise performance outcomes and serum hormonal and inflammation profiles in a cohort of young men and women.

DETAILED DESCRIPTION:
All participants were allocated to receive either gaseous hydrogen (4%) or placebo (room air) by 20-min once-per-day inhalation for 7 days, with wash-out period of 7 days to prevent the residual effects of interventions across study periods. The primary treatment outcome was the change in running time-to-exhaustion from baseline to day 7. Additionally, assessment of other exercise performance endpoints and clinical chemistry biomarkers were performed at baseline and after 7 days after each intervention.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 -35 years Body mass index 20 - 25 kg/m2 Free of major diseases Physically active Must be able to give written informed consent

Exclusion Criteria:

Use of any dietary supplements within 4 weeks before study commences Abnormal values for lab clinical chemistry (> 2 SD)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Change in exercise performance | Change from baseline running time-to-exhaustion at 7 days
  Running time-to-exhaustion

SECONDARY OUTCOMES:
Change in exercise performance | Change from baseline maximal voluntary isometric strength at 7 days
  Maximal voluntary isometric strength
Change in clinical chemistry biomarker | Change from baseline serum insulin at 7 days
  Insulin
Change in clinical chemistry biomarker | Change from baseline serum ghrelin at 7 days
  Ghrelin

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Principal Investigator — University of Novi Sad
Locations (1):
- FSPE Applied Bioenergetics Lab, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Undecided
We will provide IPD on our University repository site

REFERENCES:
- [Background] Aoki K, Nakao A, Adachi T, Matsui Y, Miyakawa S. Pilot study: Effects of drinking hydrogen-rich water on muscle fatigue caused by acute exercise in elite athletes. Med Gas Res. 2012 Jul 12;2:12. doi: 10.1186/2045-9912-2-12. eCollection 2012. PMID 22520831
- [Background] Ostojic SM. Serum alkalinization and hydrogen-rich water in healthy men. Mayo Clin Proc. 2012 May;87(5):501-2. doi: 10.1016/j.mayocp.2012.02.008. No abstract available. PMID 22560529
- [Background] Da Ponte A, Giovanelli N, Nigris D, Lazzer S. Effects of hydrogen rich water on prolonged intermittent exercise. J Sports Med Phys Fitness. 2018 May;58(5):612-621. doi: 10.23736/S0022-4707.17.06883-9. Epub 2017 Apr 26. PMID 28474871
- [Derived] Javorac D, Stajer V, Ratgeber L, Betlehem J, Ostojic S. Short-term H2 inhalation improves running performance and torso strength in healthy adults. Biol Sport. 2019 Dec;36(4):333-339. doi: 10.5114/biolsport.2019.88756. Epub 2019 Oct 31. PMID 31938004